CLINICAL TRIAL: NCT06399913
Title: Use of Cerebral Computed Tomography on Patients With Minor Head Injuries in a Danish Emergency Department: A Retrospective Cohort Study
Brief Title: Cerebral Computed Tomography on Patients With Minor Head Injuries
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: UNIFY
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Computed Tomography; Minor Head Injuries
Keywords: Emergency Department; S100B; Scandinavian Neurotrauma Committee Guideline; Traumatic Brain Injuries
MeSH Terms: conditions — Craniocerebral Trauma; Emergencies; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to calculate the prevalence of conditions or diseases requiring immediate medical attention in CTC scans with an indication of bleeding post trauma performed in the ED at Odense University Hospital. Secondary, we aim to evaluate the Scandinavian Neurotrauma Committee clinical guideline 2013 for minor head injury.

DETAILED DESCRIPTION:
In this retrospective study, our primary objectives are threefold: first, to calculate the prevalence of conditions or diseases requiring immediate medical attention and to subdivide them to explore potential correlations with biochemical, clinical, and patient baseline variables using multiple regression analysis. Secondly, we wanted to analyze our use of SNC CPG and evaluate if a more stringent application could reduce the potentially unnecessary overuse of CTC. Lastly, we aim to evaluate the 30-day mortality and readmission rates to a hospital following CTC performed in the ED.

ELIGIBILITY:
Inclusion Criteria:

* CTCs conducted from 01.01.2023 to 31.12.2023 in the ED

Exclusion Criteria:

* unrelated to trauma
* scans performed on patients under the age of 18
* CTC scans without radiologic interpretation
* Previously undergone a CTC during the same hospitalization, only the first CTC was included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CTCs conducted from 01.01.2023 to 31.12.2023 at Odense University Hospital (OUH) Emergency Department (ED) in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 7106 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Positive CTC | 1 year
  Calculate the prevalence of positive CTC findings and to subdivide them to explore potential correlations with biochemical, clinical, and patient baseline variables.
  The CT scan was acknowledged as positive if the final radiologic interpretation of all imaging studies reported one or more listed radiological findings:
  * Epidural hematoma
  * Subdural hematoma
  * Subarachnoid hematoma
  * Intraparenchymal hematoma (IPH)
  * Intraventricular hematoma
  * Fossa posterior hematoma
  * Acute infarct or dense artery sign
  * Mass effect or sulcal effacement
  * Signs of herniation
  * Basal cistern compression or midline shift
  * Cerebral contusion
  * Depressed skull fracture
  * Diastatic skull fracture
  * Pneumocephalus
  * Cerebral edema
  * Diffuse axonal injury
  * Tumor
  * Intracranial infection
  * Other which resulted in hospitalization

SECONDARY OUTCOMES:
Scandinavian Neurotrauma Committee clinical practice guideline evaluation | 1 year
  We wanted to analyze our use of SNC CPG and evaluate if a more stringent application could reduce the potentially unnecessary overuse of CTC

OTHER OUTCOMES:
30-day mortality and readmission rate | 1 year
  We aim to evaluate the 30-day mortality and readmission rates to a hospital following CTC performed in the ED.
Neurological intervention | 1 year
  The need for neurological intervention was defined as within 7 days requiring 1) neurosurgical intervention (e.g., craniotomy, hematoma evacuation, elevation of skull fracture, intracranial pressure monitoring, or intubation for head injuries indicated on CT) or 2) neuroradiological intervention (e.g., thrombectomy or intravascular embolization).

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Junghans Jensen, Principal Investigator — UNIFY, University Hospital Odense, Univeristy of Southern Denmark, OPEN
Locations (1):
- Odense University Hospital, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No